CLINICAL TRIAL: NCT00231309
Title: Pilot Study of Using Granulocyte Colony Stimulating Factor-Primed Bone Marrow in Histocompatible Sibling Allogeneic Bone Marrow Transplantation for Patients With Hematologic Malignancies and Non-Malignancies
Brief Title: Granulocyte Colony Stimulating Factor (G-CSF) for Bone Marrow Transplant (BMT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Kuang-Yueh Chiang, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0561-2003
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Hematologic Diseases; Hematologic Malignancies
Keywords: G-CSF; Bone Marrow; Hematologic malignancies; Non-malignancies; Matched sibling donor; Allogeneic BMT
MeSH Terms: conditions — Hematologic Diseases; Hematologic Neoplasms | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Other)
  Interventions: Drug: Granulocyte Colony Stimulating Factor

INTERVENTIONS:
Drug: Granulocyte Colony Stimulating Factor — Granulocyte Colony Stimulating Factor

SUMMARY:
The major purpose of this study is to evaluate the curative potential of white cell growth hormone (G-CSF)-stimulated bone marrow cells in allogeneic bone marrow transplants. Patients with cancers or blood diseases, who have poor potential for a cure with standard treatment, will be able to participate in the study. Donors will receive the white cell growth hormone (G-CSF) as a shot (injection) in their arm once a day for three days before they donate their bone marrow cells. Total body irradiation and/or chemotherapy will be given first to prepare the patient's body for the infusion of new bone marrow cells from the donor. Two medicines (cyclosporine and methotrexate) will be used to prevent the new bone marrow cells (graft) from attacking the patient's body (host) (graft-versus-host disease; GVHD). Certain safety checkpoints were built into the study if unwanted/unexpected events were to occur. If the outcomes appear better than could be expected, this will provide a bridge to extend this current approach for other innovative therapies.

DETAILED DESCRIPTION:
This study is a single-arm, non-randomized trial. Patients meeting the criteria for this study will be entered sequentially until completion or closure of the study. Early stopping rules will be employed to ascertain whether an unacceptable rate of toxicity (non-engraftment, and/or acute GvHD) occurs.

Patients will be prepared for transplant through the administration of one of the following conditioning regimen based on his/her primary disease:

5.1 Total body irradiation 1200 rads in 6 fractionated doses and high dose chemotherapy, including etoposide and cyclophosphamide.

5.2 High dose chemotherapy with busulfan and cyclophosphamide. 5.2.1 Patients who are not candidates for TBI will receive chemotherapy-based conditioning regimen.

5.3 Post transplant immunosuppression prophylaxis against acute GVHD will include cyclosporine and methotrexate.

5.4 Donor will receive 3 daily G-CSF injections (starting on day -3) prior to marrow harvest. The injections may be initiated by the donor's primary physician prior to donor's arrival here, or by BMT service at Children's Healthcare of Atlanta.

5.5 Patients will receive daily G-CSF injections (5 mcg/kg) starting from day+5 post transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancies and non-malignancies who are candidates for matched sibling donor allogeneic bone marrow transplantation are eligible for this study.
* Patients who are under 55 years of age.
* Patients who have a life expectancy of at least 12 weeks and a performance status of at least 2 Zubrod or 70% Karnofsky status prior to transplantation.
* Patients who are acceptable candidates for marrow transplantation based on their pre-BMT evaluation.
* Patients who have available histocompatible siblings who have been medically approved as marrow donors.
* Patients who sign informed consent for the protocol approved by the Institutional Review Board of Emory University/Children's Healthcare of Atlanta.
* Donors must be 5 years of age or older, and have completed routine donor evaluations and signed (by parent or legal guardian) informed consent for the protocol approved by the Institutional Review Board of Emory University/Children's Healthcare of Atlanta.

Exclusion Criteria:

* Patients will not be excluded based on sex, racial, or ethnic background.
* Patients will be excluded if they demonstrate significant functional deficits in major organs, which would obviously interfere with a successful outcome following bone marrow transplant utilizing the following guidelines:

  * Evidence of active, deep seated, life-threatening infections for which there is no known effective therapy (e.g. certain fungal species, HIV, etc.).
  * Patients with hemoglobinopathy (e.g. sickle cell disease and thalassemia) will not be eligible for this protocol. However, filgrastim mobilization, large volume apheresis, processing, and cryopreservation appears to be safe in donors with sickle cell trait.
  * Patients have had greater than two leukemic episodes, active central nervous system (CNS) and/or leukemic disease and blast crisis in chronic myelogenous leukemia (CML) patients.
* Patients will be excluded if they are women of childbearing potential who are currently pregnant (beta-hCG+) or who are not practicing adequate contraception.
* Patients who have had previous stem cell transplant will be excluded.
* Donors will be excluded if they are sensitive to E. coli-derived protein.

Max Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2003-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kuang-Yueh Chiang, M.D., Principal Investigator — Emory University/CHOA
Locations (1):
- Children's Healthcare of Atlanta/Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 patients were enrolled between July 2003 and March 2006. Patients were enrolled during consent visits for upcoming bone marrow transplants.
Pre-assignment Details: Patients were not excluded before assignment to groups.
Groups:
- Granulocyte Colony Stimulating Factor: Granulocyte Colony Stimulating Factor : Granulocyte Colony Stimulating Factor
Period: Overall Study
Arm/Group | Granulocyte Colony Stimulating Factor
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: Granulocyte Colony Stimulating Factor : Granulocyte Colony Stimulating Factor
Arm/Group | Single Arm
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.47 (4.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Participants With Disease-free Survival.
Description: Evaluate the numbers of participants with disease-free survival
Time Frame: 260 days
Measure: Number; unit: participants
Groups:
- Granulocyte-stimulating Factor: Granulocyte Colony Stimulating Factor : Granulocyte Colony Stimulating Factor
Arm/Group | Granulocyte-stimulating Factor
Number analyzed (Participants) | 10
participants | 10

2. Secondary Outcome: Hospital Length of Stay
Description: hospital length of stay of each patient enrolled, an average of 5 weeks.
Time Frame: inpatient hospital stay
Measure: Median (Standard Deviation); unit: average days
Arm/Group | Granulocyte Colony Stimulating Factor
Number analyzed (Participants) | 10
average days | 35 (70)

ADVERSE EVENTS:
Time Frame: 260 days.
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Our study is also limited by its small patient population and short follow-up time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No